CLINICAL TRIAL: NCT05789212
Title: A Personalized (N-of-1) Trial for Testing the Effect of a Mind-Body Intervention (MBI) on Sleep Duration and Quality in Middle-Aged Women Working in Healthcare
Brief Title: A Personalized Mind-Body Intervention (MBI) for Improving Sleep Among Women Working in Healthcare
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-0770; P30AG063786-01 (NIH)
Record Dates: First submitted 2023-03-13; First posted 2023-03-29 (Actual); Results first posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Sleep Insufficiency
Keywords: Sleep duration; Sleep quality; Anxiety; Depression
MeSH Terms: conditions — Sleep Deprivation; Sleep Initiation and Maintenance Disorders; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Mixed between and within (Crossover) participant assignment. The study uses a between participant randomization; each of the two arms have a multiple crossover design (with different intervention orders to the crossover).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized Trial ABCCBA (Experimental): Participants in Arm 1 will receive a Personalized Trial comprised of three components delivered in a ABCCBA sequence over a total period of 12 weeks, where A-mindfulness, B-yoga, and C-guided walking. Participants in this arm will be prompted to complete 3 x 30-minute intervention sessions weekly during applicable treatment weeks. Interventions will be delivered by a virtual link to online videos recorded by an experienced wellness provider. Participants will be limited to three views of the study-provided intervention content each week.
  Interventions: Behavioral: Personalized Trial ABCCBA
- Personalized Trial CBAABC (Experimental): Participants in Arm 2 will receive a Personalized Trial comprised of three components delivered in a CBAABC sequence over a total period of 12 weeks, where A-mindfulness, B-yoga, and C-guided walking. Participants in this arm will be prompted to complete 3 x 30-minute intervention sessions weekly during applicable treatment weeks. Interventions will be delivered by a virtual link to online videos recorded by an experienced wellness provider. Participants will be limited to three views of the study-provided intervention content each week.
  Interventions: Behavioral: Personalized Trial CBAABC

INTERVENTIONS:
Behavioral: Personalized Trial ABCCBA — Participants will receive links for 30-minute videos for all three interventions, for 2 weeks each, 3 times per week, in a specified order (ABCCBA), where A-mindfulness, B-yoga, and C-guided walking.
  Arms: Personalized Trial ABCCBA
Behavioral: Personalized Trial CBAABC — Participants will receive links for 30-minute videos for all three interventions, for 2 weeks each, 3 times per week, in a specified order (CBAABC), where A-mindfulness, B-yoga, and C-guided walking.
  Arms: Personalized Trial CBAABC

SUMMARY:
The goal of this pilot study is to determine if a personalized trial testing a Mind-Body Intervention (MBI) can produce a meaningful increase in the average daily sleep duration among women 40-60 years of age working in healthcare. A total of 60 eligible participants will be randomized to one of two possible orders of treatment exposure comprised of three components: mindfulness, yoga, and guided walking, each assigned in 2-week block sequences for a total period of 12 weeks. The study will include a 2-week baseline period during which their baseline sleep duration and adherence to the Fitbit wear and survey submission will be assessed. Following the 2-week run-in period, participants deemed eligible and achieved at least 80% adherence of Fitbit wear and survey submission will be randomized to one of the two intervention arms. Exploratory aims include assessments of sleep quality, physiological factors and their direct and indirect relationships with participants' perceived stress, anxiety, and depression.

DETAILED DESCRIPTION:
The goal of this pilot study is to determine if a personalized trial (N-of-1) employing a Mind-Body Intervention (MBI) can produce a meaningful increase in sleep duration among women 40-60 years of age working at Northwell Health. A total of 60 women with a history of short sleep duration (defined as an average <7h per 24-h period for at least three months) will be enrolled over a period of two years. Participants will complete a 2-week run-in period with no intervention, during which their baseline sleep duration and adherence to the Fitbit wear and survey submission will be assessed. Adherence to Fitbit wear will be defined as recorded activity of greater than 12 hours a day, and recorded sleeping activity greater than 180 minutes in total. Survey adherence will be defined as submission of a given survey. Participants who achieve at least 80% adherence of Fitbit wear and survey submission during baseline period will be randomized to Arm 1 (N=30) or Arm 2 (N=30). Each arm will receive a personalized intervention comprised of three components: mindfulness, yoga and guided walking assigned in 2-week block sequences for a total period of 12 weeks. During each 2-week block, participants will be prompted to complete 3 x 30-minute intervention sessions weekly. Interventions will be delivered by a virtual link to online videos recorded by an experienced wellness provider. Participants will be limited to three views of the study-provided intervention content each week. Changes in average daily sleep duration will be calculated for each participant based on daily measurements between the run-in and each treatment period. The Fitbit devices will also record sleep quality components (sleep onset, sleep staging, and overall sleep score) and physiological factors (breathing/resting heart rate, heart rate variability (HRV) and activity). We will also examine the direct and indirect relationships between perceived stress, anxiety and depression, and sleep quality assessed pre, during (bi-weekly), and post MBI. Enrollment will continue until up to 60 participants have been randomized. Following the intervention, all participants will be assessed over a 2-week follow-up period to allow for a personalized report of their observed data to be generated.

ELIGIBILITY:
Inclusion Criteria:

* Women (biological sex at birth)
* Age 40-60 years old
* Northwell employee/affiliate
* Self-reported history of short sleep duration (<7h per 24-h period) for at least 3 months
* After 2-week run-in, Fitbit-verified short sleep duration and ≥80% adherence of Fitbit wear and survey submission
* Self-report of perceived stress ≥18 using the Perceived Stress Scale (PSS)
* Access to and capable of using a smartphone
* Can regularly wear a Fitbit device

Exclusion Criteria:

* Men (biological sex at birth)
* Age < 40 or >60 years old
* Women who are pregnant
* Not a Northwell employee/affiliate
* No history of short sleep duration or non-adherent to the Fitbit wear and survey submission
* Self-report of perceived stress <18 using the Perceived Stress Scale (PSS)
* Does not own or cannot regularly access a smartphone
* Cannot regularly wear a Fitbit device
* Unable to complete the study due to cognitive impairment, severe medical or mental illness, or active/prior substance abuse
* Planned surgeries 6 months from study start date
* Participants who have been previously told by a doctor/clinician they have mobility limiting health conditions and/or to not engage in walking 30 minutes, three times per week or yoga

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2025-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karina Davidson, PhD, MASc, Principal Investigator — Northwell Health
Locations (1):
- Institute of Health System Science, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participant data (IPD) will be de-identified and pooled before sharing on the Open Science Framework, along with a data dictionary.
Supporting Information: Study Protocol, SAP
Time Frame: The study protocol, including the statistical analysis plan, will be made available in addition to the informed consent form following completion of recruitment but prior to publication of any data from the current study. De-identified, pooled individual participant data will be made available within a year of final participant data collection. We anticipate this data to be available on the Open Science Framework platform indefinitely.
Access Criteria: All data and supporting information will be stored on the Open Science Framework, a free web application with no access restrictions.

RESULTS

PARTICIPANT FLOW:
Groups:
- Personalized Trial Group 1 (ABCCBA): Participants in Arm 1 will receive a Personalized Trial comprised of three components delivered in a ABCCBA sequence over a total period of 12 weeks, where A-mindfulness, B-yoga, and C-guided walking. Participants in this arm will be prompted to complete 3 x 30-minute intervention sessions weekly during applicable treatment weeks. Interventions will be delivered by a virtual link to online videos recorded by an experienced wellness provider. Participants will be limited to three views of the study-provided intervention content each week.
  Personalized Trial ABCCBA: Participants will receive links for 30-minute videos for all three interventions, for 2 weeks each, 3 times per week, in a specified order (ABCCBA), where A-mindfulness, B-yoga, and C-guided walking.
- Personalized Trial Group 2 (CBAABC): Participants in Arm 2 will receive a Personalized Trial comprised of three components delivered in a CBAABC sequence over a total period of 12 weeks, where A-mindfulness, B-yoga, and C-guided walking. Participants in this arm will be prompted to complete 3 x 30-minute intervention sessions weekly during applicable treatment weeks. Interventions will be delivered by a virtual link to online videos recorded by an experienced wellness provider. Participants will be limited to three views of the study-provided intervention content each week.
  Personalized Trial CBAABC: Participants will receive links for 30-minute videos for all three interventions, for 2 weeks each, 3 times per week, in a specified order (CBAABC), where A-mindfulness, B-yoga, and C-guided walking.
Period: Overall Study
Arm/Group | Personalized Trial Group 1 (ABCCBA) | Personalized Trial Group 2 (CBAABC)
Started | 30 | 30
First Intervention Block (2 Weeks) | 30 | 30
Second Intervention Block (2 Weeks) | 30 | 29
Third Intervention Block (2 Weeks) | 30 | 29
Fourth Intervention Block (2 Weeks) | 29 | 28
Fifth Intervention Block (2 Weeks) | 29 | 28
Sixth Intervention Block (2 Weeks) | 29 | 28
Follow-Up Block (2 Weeks) | 29 | 28
Completed | 29 | 27
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Personalized Trial Group 1 (ABCCBA) | Personalized Trial Group 2 (CBAABC) | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.53 (5.98) | 49.20 (6.69) | 48.87 (6.30)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 26 | 25 | 51
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 4 | 10
  White | 14 | 19 | 33
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Mean Within-Subject Difference in Daily Sleep Duration
Description: The effect of the personalized MBI intervention on individual's sleep duration will be assessed in each arm separately. Participants' daily sleep duration will be measured objectively using Fitbit devices and by self-reported questionnaires. Individual changes in the average daily sleep durations between the run-in and each treatment period will be reported using means and 95% CIs. Bland-Altman plots will be constructed to visualize agreement between Fitbit reported and self-reported sleep duration. The effects of treatment on sleep duration will be assessed using GEE with an unstructured variance-covariance matrix for measures on the same day to that night's sleep. This model accounts for possible autocorrelation and linear trends between sleep duration across time.
  A change between time points is reported (e.g., baseline (2 weeks) and 2 weeks for each intervention period (4 weeks per intervention)) as a value for each intervention period minus value at baseline.
Time Frame: Baseline (2 weeks) and 2 weeks for each intervention period (4 weeks total for each intervention)
Measure: Mean (95% Confidence Interval); unit: minutes per day
Groups:
- Overall (All Participants): Participants in Arm 1 and Arm 2
Arm/Group | Personalized Trial Group 1 (ABCCBA) | Personalized Trial Group 2 (CBAABC) | Overall (All Participants)
Number analyzed (Participants) | 30 | 30 | 60
minutes per day
  Guided Walking (C) | 0.10 [-12.6 to 12.8] | 3.45 [-12.0 to 18.9] | 1.74 [-7.04 to 10.5]
  Mindfulness Meditation (A) | 0.43 [-11.9 to 12.8] | 1.66 [-14.1 to 17.4] | 0.81 [-7.94 to 9.57]
  Yoga (B) | -2.89 [-15.2 to 9.41] | 5.94 [-9.78 to 21.7] | 1.27 [-7.43 to 9.97]

2. Other Pre Specified Outcome: Mean Within-Subject Difference in Daily Sleep Latency
Description: Sleep latency is an important parameter in a sleep study. The duration of time between when the lights are turned off (lights out) as the patient attempts to sleep, until the time patient actually falls asleep will be reported as sleep latency and aggregated daily using Fitbit devices. The effect of the personalized MBI intervention on individual's sleep latency will be assessed in each arm separately. Individual changes in the average daily sleep latency between the run-in and each treatment period will be reported using means (95% CIs) and modeled using Generalized estimating equations (GEE).
Time Frame: 13-16 weeks
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Mean Within-Subject Difference in Daily Sleep Efficiency
Description: Sleep efficiency (SE) is an indicator of sleep quality. SE is commonly defined as the ratio of total sleep time (TST) to time in bed (TIB). Values (as percentages) greater than or equal to 85% indicate good sleep quality (Ohayon et al., 2017 [PMID: 28346153]). SE will be recorded and aggregated daily using Fitbit devices. The effect of the personalized MBI intervention on individual's SE be assessed in each arm separately. Individual changes in the average daily sleep efficiency between the run-in and each treatment period will be reported using means (95% CIs) and modeled using Generalized estimating equations (GEE).
Time Frame: 13-16 weeks
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Mean Within-Subject Difference in Daily Resting Heart Rate
Description: Fitbit calculates the resting heart rate by measuring the heart rate when it detects sleep, and by measuring it throughout the day while an individual is but inactive (no steps detected). Resting heart rate will be recorded and aggregated daily using Fitbit devices. The effect of the personalized MBI intervention on individual's resting heart rate will be assessed in each arm separately. Individual changes in the average resting heart rate between the run-in and each treatment period will be reported using means (95% CIs) and modeled using Generalized estimating equations (GEE).
Time Frame: 13-16 weeks
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Mean Within-Subject Difference in Daily Number of Steps
Description: The number of steps per day (physical activity) will be recorded and aggregated daily using Fitbit devices. The effect of the personalized MBI intervention on individual's number of steps per day will be assessed in each arm separately. Individual changes in the daily average number of steps between the run-in and each treatment period will be reported using means (95% CIs) and modeled using Generalized estimating equations (GEE).
Time Frame: 13-16 weeks
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Mean Within-Subject Difference in Perceived Stress Score
Description: Participant's perceived stress score will be measured using the Perceived Stress Scale (PSS) (scale 0 to 40) and the Ecological Momentary Assessment (EMA) Stress questionnaire (scale 0 to 10). PSS and EMA will be evaluated pre-intervention (run-in), bi-weekly during the intervention, and post-intervention. Individual changes in the average PSS and EMA scores between the run-in and each treatment period will be reported using means (95% CIs).
Time Frame: 13-16 weeks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Mean Within-Subject Difference in Anxiety and Depression Scores
Description: Participant's anxiety and depressive disorder scores will be assessed using the Patient Health Questionnaire (PHQ-4), a self-report version of the Primary Care Evaluation of Mental Disorders (PRIME-MD) on a scale of 0 to 3 for a total of four items. Total score will be determined by adding together the scores of each of the 4 items. Scores are rated as normal (0-2), mild (3-5), moderate (6-8), and severe (9-12). Total score ≥3 for first 2 questions suggests anxiety. Total score ≥3 for last 2 questions suggests depression. PHQ-4 will be evaluated pre-intervention (run-in), bi-weekly during the intervention, and post-intervention. Individual changes in the average PHQ-4 scores between the run-in and each treatment period will be reported using means (95% CIs). The role of anxiety and depression as a potential mediator (M) between perceived stress (X) and sleep score (Y), will be determined by mixed effects regression models.
Time Frame: 13-16 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Non-systematic adverse event data was collected over the course of the 16-week trial: 2-week baseline period, 12-week intervention, and 2-week follow-up period.
Groups:
- Mindfulness Meditation (A): Mindfulness meditation (Intervention A) was delivered to participants in the Personalized Trials arms as part of their ABCCBA and CBAABC intervention sequences. Participants were asked to complete virtual mindfulness meditation sessions via link to an online video 3 times per week in 2-week blocks.
- Yoga (B): Yoga (Intervention B) was delivered to participants in the Personalized Trials arms as part of their ABCCBA and CBAABC intervention sequences. Participants were asked to complete virtual yoga sessions via link to an online video 3 times per week in 2-week blocks.
- Walking (C): Walking (Intervention C) was delivered to participants in the Personalized Trials arms as part of their ABCCBA and CBAABC intervention sequences. Participants were asked to complete virtual walking sessions via link to an online video 3 times per week in 2-week blocks.
- No Intervention (Baseline): The 2-week baseline period at the start of the trial to determine eligibility for the intervention period. No interventions delivered during baseline.
Arm/Group | Mindfulness Meditation (A) | Yoga (B) | Walking (C) | No Intervention (Baseline)
All-Cause Mortality (participants affected / at risk) | 4/60 | 1/60 | 2/60 | 5/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60 | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 3/60 | 0/60 | 2/60 | 1/60
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mindfulness Meditation (A) (N=60) | Yoga (B) (N=60) | Walking (C) (N=60) | No Intervention (Baseline) (N=60)
Skin irritation from Fitbit device (General disorders) | 3 (3) | 0 (0) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-26): https://cdn.clinicaltrials.gov/large-docs/12/NCT05789212/Prot_SAP_001.pdf
  • Informed Consent Form (2023-10-26): https://cdn.clinicaltrials.gov/large-docs/12/NCT05789212/ICF_000.pdf